CLINICAL TRIAL: NCT07066748
Title: Weaning From Mechanical Ventilation After Pediatric Cardiac Surgery. A Randomized Controlled Trial
Brief Title: Weaning From Mechanical Ventilation After Pediatric Cardiac Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Islam Elbardan, LECTURER OF ANESTHESIA AND SURGICALMINTENSIVE CARE, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: serial number:0307330
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Weaning Mechanical Ventilation; Pediatric Cardiac Surgery
Keywords: automatic tube compensation; congenital cardiac anomalies
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P: weaning using pressure support ventilation mode (Active Comparator): Group P: Weaning trial will be done for patients using PSV 8 cmH2O without ATC.
  Interventions: Procedure: group P:pressure support ventilation mode
- group A:Autmated tube compensation mode (Experimental): Group A: Weaning trial will be done for patients using PSV 0 cmH2O with 100% automatic tube compensation (ATC).
  Interventions: Procedure: group A:automatic tube compensation (ATC).

INTERVENTIONS:
Procedure: group P:pressure support ventilation mode — Group P: Weaning trial will be done for patients using PSV 8 cmH2O without ATC
  Arms: Group P: weaning using pressure support ventilation mode
Procedure: group A:automatic tube compensation (ATC). — Group A: Weaning trial will be done for patients using PSV 0 cmH2O with 100% automatic tube compensation (ATC).
  Arms: group A:Autmated tube compensation mode

SUMMARY:
Weaning from mechanical ventilation post congenital cardiac surgery is often challenging. It is well known that not all patients can be early extubated, although most are suitable for early postoperative weaning and extubating despite complex operative procedures. With advances in anaesthesia management, cardiopulmonary bypass (CPB), and surgical techniques, the trend of 'fast tracking', and early extubating of pediatrics postcardiac surgery seems to be feasible. Unnecessary prolonged mechanical ventilation increases the complication risks as airway trauma, ventilator associated pneumonia, and increased hospital stay

DETAILED DESCRIPTION:
Different methods have been used to predict the optimum time to make the weaning decision. These methods include, success of spontaneous breathing trials (SBTs), counting respiratory rate, observation of work of breathing, and many other calculated indices such as hypoxic index, oxygenation index, stress index, oxygen reserve index, dynamic compliance, and rapid shallow breathing index (RSBI). However, some of these indices may be misleading and not precise.

Pressure support ventilation (PSV) has been widely used in the performance of a spontaneous breathing trial because it can compensate to some extent for the additional work of breathing imposed by the endotracheal tube and the breathing circuit. However, it is difficult to recognize the exact pressure support to overcome the tubing resistance during the weaning process till extubating.

The ventilator modality of automatic tube compensation (ATC) can provide variable pressure supports during the weaning process to overcome any change in the resistance of the breathing circuit, endotracheal tube, and airways. ATC is effective in overcoming the work of breathing caused by airway resistance to allow successful weaning process and extubating.

Several studies have investigated the effectiveness of ATC and PS for ventilatory weaning in adult patients, with conflicting results. Fewer studies have focused on the pediatric population, and even fewer have specifically examined patients who have undergone cardiac surgery. Therefore, there is a need for further research to determine the most effective weaning mode for this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2-10years.
2. Both sex.
3. after fulfilling weaning criteria
4. being pain free (observational pain/discomfort scale < 4). the weaning criteria; which include: low mandatory ventilator rate [6-8] or less; fraction of inspired oxygen (FIO2) ≤ 40; level of positive end expiratory pressure (PEEP) [3-5 cmH2O] guided by pressure/volume loop; reversal of the cause of postoperative mechanical ventilation; oxygenation index (OI) (mean air way pressure × FIO2/PaO2) < 5; dynamic compliance (Cdyn) > 1 ml/ cmH2O/kg

Exclusion Criteria:

1. Duration of mechanical ventilation is more than 48 hours
2. Patients on high inotropic support (unstable hemodynamics)
3. Patients with disturbed conscious level
4. Patients with palliative cardiac shunting procedures (e.g., BT shunt, Glenn shunt).

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
work of breathing (WOB) | during weaning trial 30 minutes
  compare the efficacy of ATC versus PS as a modality for ventilatory weaning of pediatric postcardiac surgery as regards effects on work of breathing, (WOB) (∆ V × flow × R + Volume/compliance) (J/L/Kg).
lung compliance | during ventilatory weaning in 30 minutes
  to compare the efficacy of ATC versus PS as a modality for ventilatory weaning of pediatric postcardiac surgery as regards effects on lung compliance. Dynamic compliance (Cdyn) (ml/cmH2O/kg).
alveolar recruitment | base line immediately before starting weaning trial, every 15 minutes during the weaning trial and 15 minutes after extubating
  by Ultrasound lung aeration score: assessment of the lung atelectasis by the lung ultrasound examination, six basic regions will be assessed for each lung. Each hemithorax is divided into anterior, lateral and posterior regions by the anterior and posterior axillary lines. The regions are further subdivided into upper and lower areas. Characteristics Points Normal aeration or less than 2 isolated B lines 0 Moderate loss of aeration with multiple, well-defined B-lines 1 Severe loss of aeration with multiple coalescent B-lines 2 Lung consolidation 3

SECONDARY OUTCOMES:
Numbers of weaning trials. | 48 hour post operative
recording the requirement for reintubation and mechanical ventilation | within 48 hours after extubation
  Requirement for reintubation and mechanical ventilation after prior successful weaning from ventilation,

CONTACTS AND LOCATIONS:
Overall Officials: LECTURER OF ANESTHESIA AND SURGICAL INTENSIVE CARE, Dr, Principal Investigator — University of Alexandria
Locations (1):
- Faculty of medicine ,Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No